CLINICAL TRIAL: NCT06942611
Title: A Study on the Therapeutic Effects of Transcranial Electrical Stimulation Combined on Chronic Pain in Central Nervous System Inflammatory Demyelinating Diseases
Brief Title: Transcranial Electrical Stimulation for Treating Chronic Pain in Inflammatory Demyelinating Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: xw-tES-03
Record Dates: First submitted 2025-01-19; First posted 2025-04-24 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Inflammatory Demyelinating Disorders of the Central Nervous System

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurostimulation group (Experimental)
  Interventions: Device: transcranial electrical stimulation treatment.
- Sham neurostimulation group (No Intervention)

INTERVENTIONS:
Device: transcranial electrical stimulation treatment. — Stimulation targeting the primary motor cortex, current intensity is 1-2mA, duration is 30 minutes, once daily for 5 consecutive days
  Arms: Neurostimulation group

SUMMARY:
Non-invasive neurostimulation can effectively improve patients' symptoms and has shown good therapeutic efficacy in alleviating the symptoms of IIDDs (Inflammatory Immune-mediated Demyelinating Diseases). However, some patients have not achieved the desired results, which may be due to individual differences in neural responsiveness . Therefore, this study aims to assess the therapeutic effect of transcranial electrical stimulation on improving symptoms such as painful spasm in IIDDs patients, by considering both the overall characteristics of IIDDs disease symptoms and individual differences in patients. The study will explore the imaging characteristics, electrophysiological features of the disease symptoms, and their relationship with clinical manifestations, while analyzing the key factors that influence treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with neuromyelitis optica spectrum disorder, multiple sclerosis, or other central nervous system inflammatory demyelinating diseases that meet the diagnostic criteria;

Numeric Rating Scale (NRS) pain score ≥4;

Age between 18 and 65 years, regardless of gender;

Stable dose of immunosuppressive therapy for at least one month;

EDSS score ≤6;

Right-handed;

Agree to participate and sign the informed consent form.

Exclusion Criteria:

A history of relapse within the past month;

Recent medication adjustments or treatment with modified electroconvulsive therapy, transcranial magnetic stimulation, or other neurostimulation techniques within the past month;

Participation in any other clinical trial within the past month or currently participating in another clinical trial;

Presence of cochlear implants, pacemakers, or implanted stimulators in the brain;

Skin integrity at the electrode placement site is compromised, or allergy to electrode gel or adhesive;

A history of epilepsy, hydrocephalus, central nervous system tumors, brain injury, or intracranial infections;

Pregnant or breastfeeding women, or those planning to become pregnant in the near future;

A score of ≥3 on item 3 (suicide item) of the HDRS-17, or a history of severe psychiatric disorders;

Presence of severe or unstable organic diseases;

Poor patient compliance preventing cooperation with treatment, follow-up, or clinical, EEG, and imaging data collection;

Any other situation deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-03 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | From enrollment to the end of treatment at 1 month
  VAS Score (Visual Analog Scale) is a commonly used tool to assess pain intensity. It usually consists of a line marked with "no pain" (0 points) and "worst possible pain" (such as 0-100 points). The patient marks their level of pain on the line to provide a score. The advantage of the VAS is its simplicity, clarity, and ease of use for patients.

SECONDARY OUTCOMES:
NRS scores | From enrollment to the end of treatment at 1 month
  The NRS (Numerical Rating Scale) is a self-reported tool that measures pain intensity on a scale from 0, indicating no pain, to 10, representing the worst possible pain.
SF-MPQ scores | From enrollment to the end of treatment at 1 month
  The SF-MPQ (Short-Form McGill Pain Questionnaire) measures pain quality and intensity using a set of descriptive words rated on an intensity scale; higher scores indicate greater pain severity.
Modified Ashworth scale | From enrollment to the end of treatment at 1 month
  The Modified Ashworth Scale (MAS) is used to assess muscle spasticity by measuring resistance during passive soft-tissue stretching, with scores ranging from 0 (no increase in muscle tone) to 4 (rigid in flexion or extension), where higher scores indicate greater spasticity.
The HAMD (Hamilton Depression Rating Scale) scores | From enrollment to the end of treatment at 1 month
  The HAMD (Hamilton Depression Rating Scale) is a clinician-administered questionnaire used to assess the severity of depression, with scores typically ranging from 0 to 52; higher scores indicate more severe depressive symptoms.
The HAMD (Hamilton Anxiety Rating Scale) scores | From enrollment to the end of treatment at 1 month
  The HAMD Anxiety Subscale refers to the anxiety-related items within the Hamilton Depression Rating Scale, which are used to assess both psychological and somatic symptoms of anxiety, such as tension, worry, restlessness, fear, and somatic complaints. Higher scores indicate more severe anxiety symptoms. This subscale is clinician-rated and commonly used to evaluate anxiety levels in patients with depression.
Fatigue Severity Scale | From enrollment to the end of treatment at 1 month
  The FSS (Fatigue Severity Scale) is a self-reported questionnaire used to assess the impact of fatigue on a person's daily functioning, consisting of 9 items rated on a scale from 1 (strongly disagree) to 7 (strongly agree); higher scores indicate more severe fatigue.
MMSE (Mini-Mental State Examination) Score | From enrollment to the end of treatment at 1 month
  The MMSE (Mini-Mental State Examination) is a widely used clinician-administered tool for screening cognitive function, with scores ranging from 0 to 30; higher scores indicate better cognitive performance, while lower scores suggest cognitive impairment.
Epworth Sleepiness Scale scores | From enrollment to the end of treatment at 1 month
  The ESS (Epworth Sleepiness Scale) is a self-reported questionnaire used to assess daytime sleepiness by asking individuals to rate their likelihood of dozing off in various daily situations; scores range from 0 to 24, with higher scores indicating greater daytime sleepiness.
Short Form Health Survey-36 Score | From enrollment to the end of treatment at 1 month
  The SF-36 (Short Form Health Survey-36) is a self-reported questionnaire that measures overall health-related quality of life across eight domains, including physical functioning, bodily pain, general health, and mental health. Scores for each domain range from 0 to 100, with higher scores indicating better health status and quality of life.
EEG features of Absolute Power | From enrollment to the end of treatment at 1 month
  Reflects the raw amplitude strength within a specific frequency band (e.g., delta, theta, alpha, beta, gamma), calculated by integrating the power spectral density (PSD) over that band.
EEG features of Absolute Power | From enrollment to the end of treatment at 1 month
  Power spectral analysis of EEG data quantifies the distribution of signal power across different frequency bands(e.g., delta, theta, alpha, beta, gamma), providing insights into the brain's oscillatory activity. It is typically performed using Fourier or wavelet transforms to compute.
Functional Connectivity of EEG data | From enrollment to the end of treatment at 1 month
  the statistical dependencies between spatially separated brain regions, reflecting how different parts of the brain communicate during rest.
Microstate Analysis of EEG data | From enrollment to the end of treatment at 1 month
  EEG microstate analysis involves segmenting the continuous EEG signal into short periods of quasi-stable topographic maps, each representing a distinct brain functional state. These microstates are identified using clustering algorithms (e.g., k-means) on scalp voltage maps derived from the EEG's global field power peaks.
Nonlinear Dynamics of EEG data | From enrollment to the end of treatment at 1 month
  Nonlinear dynamics of EEG data provide a general measure of the brain's complexity and the unpredictable nature of neural activity. These analyses help reveal hidden patterns and dynamic properties that are not captured by traditional linear methods.
Graph theory metrics of EEG data | From enrollment to the end of treatment at 1 month
  Graph theory metrics of EEG data characterize the brain's functional network organization by modeling connectivity patterns as a graph of nodes (electrodes or regions) and edges (functional connections).
Structural measures from T1-weighted MRI | From enrollment to the end of treatment at 1 month
  Structural measures from T1-weighted MRI assess the brain's anatomical properties
Functional measures of resting-state fMRI | From enrollment to the end of treatment at 1 month
  Functional measures of resting-state fMRI capture spontaneous brain activity and inter-regional communication by analyzing low-frequency BOLD signal fluctuations.
The Pittsburgh Sleep Quality Index (PSQI) | From enrollment to the end of treatment at 1 month
  The Pittsburgh Sleep Quality Index (PSQI) is a self-administered questionnaire that assesses subjective sleep quality and disturbances over a one-month period. It generates seven component scores (including sleep latency, duration, efficiency and disturbances) which are summed into a global score (0-21), with higher scores indicating poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No